CLINICAL TRIAL: NCT00934713
Title: The Effect of Montelukast Therapy on Respiratory Symptoms, Lung Function and Airway Responsiveness in Wheezy Very Young Children
Brief Title: The Effect of Montelukast Treatment in Wheezy Infants
Acronym: Montelukast
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Pelkonen Anna, Helsinki University Central Hospital, P.O.Box 160, FIN-00029, Finland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 33902
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2003-10

CONDITIONS: Lung Disease, Obstructive; Signs and Symptoms, Respiratory
Keywords: montelukast, very young children, lung function tests
MeSH Terms: conditions — Lung Diseases, Obstructive; Signs and Symptoms, Respiratory | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- montelukast (Active Comparator): montelukast 4 mg once per day for 8 weeks
  Interventions: Drug: montelukast

INTERVENTIONS:
Drug: montelukast — montelukast 4mg once per day for 8 weeks period
  Other Names: singulair

SUMMARY:
The study is designed to evaluate the efficacy of montelukast on symptom-free days in unselected group of very young children with wheeze and recurrent asthma like symptoms. The secondary aim was to evaluate the effect of montelukast on lung function, airway responsiveness, airway inflammation and use of rescue medication.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effectiveness of montelukast in wheezy very young children with persistent respiratory symptoms. This study was a prospective, double-blind, placebo-controlled study of 6 to 24 months old children, who had at least one physician-diagnosed wheezing episode and persistent asthmatic symptoms. Patients were randomised to placebo or montelukast 4 mg / day for 8 weeks period. The clinical response to treatment was determined, the functional residual capacity (FRC) and specific air-way conductance (sGaw) was measured using an infant whole-body pletys-mograph, the maximal flow at functional residual capacity (V´maxFRC) was re-corded using the squeeze technique and airway responsiveness was evaluated by performing a dosimetric methacholine challenge test.

ELIGIBILITY:
Inclusion Criteria:

* at least one physician-diagnosed wheezing episode and history of recurrent cough, dyspnoea and wheeze and successfully performed methacholine challenge test were included.

Exclusion Criteria:

* use of ICS within 8 weeks prior to the first visit, a cumulative life-time systemic prednisolone use more than 3 days at a dose of 2 mg/kg, an equipotent dose of another systemic corticosteroid or ICS use more than 4 weeks, respiratory infection in the 14 days preceding lung function measurement and obvious tracheobronchomalacia or other structural defect.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2004-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
symptom free days | 2 weeks runin and 8 weeks treatment

SECONDARY OUTCOMES:
lung function, airway responsiveness, exhale nitric oxide, use of rescue medication | before and after 8 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anna S Pelkonen, MD, Study Chair — Helsinki University Central Hospital
Locations (1):
- Skin and Allergy Hospital, Helsinki University Central Hospital, Helsinki, P.O.Box 160, Finland

REFERENCES:
- [Derived] Pelkonen AS, Malmstrom K, Sarna S, Kajosaari M, Klemola T, Malmberg LP, Makela MJ. The effect of montelukast on respiratory symptoms and lung function in wheezy infants. Eur Respir J. 2013 Mar;41(3):664-70. doi: 10.1183/09031936.00173411. Epub 2012 Jul 12. PMID 23060628